CLINICAL TRIAL: NCT01461278
Title: A Prospective, Randomized, Single-Masked, Controlled, Parallel Groups, Multicenter Clinical Investigation of the Glaukos® Suprachoroidal Stent Model G3 In Conjunction With Cataract Surgery
Brief Title: Multicenter Investigation of the Glaukos® Suprachoroidal Stent Model G3 In Conjunction With Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GC-007
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Primary open-angle glaucoma; POAG; Cataract surgery; Suprachoroidal space; Suprachoroidal stent; iStent supra
MeSH Terms: conditions — Glaucoma, Open-Angle; Choroidal Effusions | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cataract surgery plus iStent supra (Experimental)
  Interventions: Device: iStent supra; Procedure: Cataract surgery
- Cataract surgery (Active Comparator)
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Device: iStent supra — Cataract surgery and implantation of one iStent supra
  Arms: Cataract surgery plus iStent supra
Procedure: Cataract surgery — Cataract surgery alone

SUMMARY:
Evaluate the safety and efficacy of the Glaukos® Suprachoroidal Stent Model G3 in conjunction with cataract surgery, compared to cataract surgery only, in subjects with mild to moderate primary open-angle glaucoma.

DETAILED DESCRIPTION:
This is an IDE trial to evaluate the safety and efficacy of the Glaukos® Suprachoroidal Stent Model G3 (hereinafter referred to as G3) in conjunction with cataract surgery, compared to cataract surgery only, in subjects with mild to moderate primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate open-angle glaucoma
* Characteristics consistent with mild to moderate glaucoma
* Use of one (1) to three (3) medications at time of screening exam

Exclusion Criteria:

* Pigmentary or pseudoexfoliative glaucoma
* Prior incisional glaucoma surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2011-12-22 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
≥ 20% Reduction in Intraocular Pressure (IOP) | Baseline and Month 24

SECONDARY OUTCOMES:
Diurnal IOP Reduction from Baseline | Baseline and Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, O.D., Study Chair — Glaukos Corporation
Locations (1):
- Eye Centers of Racine and Kenosha, Racine, Wisconsin, United States